CLINICAL TRIAL: NCT06240052
Title: Use Electroencephalogram to Study Neural Dynamics of Fear Conditioning and Avoidance Learning Circuit in Humans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mohammed Milad, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-23-0841
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Neural Dynamics of the Acquisition and Retention of Fear Learning and Active Avoidance Learning
Keywords: Fear Learning; Active Avoidance; Electroencephalogram (EEG)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conditioning and active avoidance paradigm (CAAP) (Experimental)
  Interventions: Behavioral: Conditioning and active avoidance paradigm (CAAP)

INTERVENTIONS:
Behavioral: Conditioning and active avoidance paradigm (CAAP) — On day 1 subjects will undergo image viewing, fear conditioning, and avoidance learning. Subjects will be instructed to passively view the images from 3 categories on the screen, with 2 of the 3 categories being paired with a mild shock to the subjects' foot. Then they will see a picture of a button on the screen together with all three categories. If they press the button, they may prevent the shock from occurring. Pressing the button for one of the conditioned categories will prevent the shock from happening. Pressing the button to the other conditioned cue will not prevent the shock .Pressing the button to the third category does nothing. On day 2, subjects will be given $5 and will be told that they can press a button to avoid a shock. The number of times the button was pressed will be counted and if it is less than the number by another randomly selected participant then the participant will get to keep the money.

SUMMARY:
The purpose of this study is to examine which event-related potentials (ERPs) and event-related oscillations (EROs) are associated with fear conditioning, avoidance learning, and memory recall for fear and avoidance, where are the source generators of the observed scalp EEG activity, the impact of fear and avoidance learning on the decision to avoid or not to avoid conditioned stimuli , to examine the large-scale functional connectivity across distributed brain regions across experimental phases, and to examine whether spontaneous EEG data during resting-state correlate with the EEG measures during experimental tasks.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent.

Exclusion Criteria:

* History of neurologic disease
* History of seizure or significant head trauma/loss of consciousness
* Significant serious psychiatric diagnosis
* Significant suicidal ideation or behaviors
* High risk of adverse emotional or behavioral reaction, and/or an inability to understand study procedures or the informed consent process, based on investigator/clinician clinical evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Skin Conductance Response (SCR) during the image familiarization phase (viewing phase) | During the image familiarization/viewing phase (about 15 minutes total)
  On day 1 during the image familiarization phase (also called the viewing phase), participants will be presented with images on a computer screen from three different object categories, such as fruits, animals, and tools, and participants will be instructed to passively view the presented images.
  During the viewing phase, Skin Conductance Response (SCR) will be recorded to assess participants' response to each object category. SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each of the 3 object categories.
Skin Conductance Response (SCR) during the fear conditioning phase | During the fear conditioning phase (about 18 minutes total)
  In this phase participants will continue to be presented with images from the three categories, which will be used as conditioned stimuli (CS), as follows. Objects from two categories will be reinforced by a mild electrical shock (CS+), whereas the third category will never be reinforced (CS-). Skin Conductance Response (SCR) will be recorded to assess participants' response to each object category. SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated. SCR will be reported in microsiemens for each of the 3 object categories.
Skin Conductance Response (SCR) during the avoidance learning phase | During the avoidance learning phase (about 18 minutes total)
  On day 1, after the fear phase, participants will complete the avoidance learning phase. In this phase, participants can avoid a shock by pressing a button. Objects from some categories will be reinforced by a mild electrical shock (CS+), whereas the other categories will not be reinforced (CS-). Pressing the button during the presentation of the object will or will not prevent the shock from occurring. During the avoidance learning phase, Skin Conductance Response (SCR) will be recorded to assess participants' response to each object category. SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each of the 3 object categories.
Skin Conductance Response (SCR) during the memory recall phase | During the memory recall phase (about 18 minutes total)
  On day 2, participants will complete the memory recall phase. During this phase, participants will again be presented with images on a computer screen from three different object categories, such as fruits, animals, and tools. Participants will be informed that they have a choice to press or not to press a button during the image presentation to avoid a possible shock.
  During the memory recall phase, Skin Conductance Response (SCR) will be recorded to assess participants' response to each object category. SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each of the 3 object categories.
Skin Conductance Response (SCR) during resting state | Immediately Before the Viewing Phase on day 1
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately After the Viewing Phase (day 1 about 15 minutes after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately Before the fear conditioning Phase (day 1 about 20 minutes after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately After the fear conditioning Phase (day 1 about 38 minutes after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2). SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately Before the avoidance learning phase (day 1 about 43 minutes after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately after the avoidance learning phase (day 1 about 61 minutes after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately Before the memory recall phase on day 2 (about 1 day after start of viewing phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
  SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Skin Conductance Response (SCR) during resting state | Immediately after the memory recall phase (day 2 about 1 day 18 minutes after start of memory recall phase)
  Skin Conductance Response (SCR) in microsiemens will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2). SCR is measured by placing two electrodes on the skin and passing a tiny electric charge between the two points. SCR is proportionally related to the number of sweat glands that are activated, meaning that the more emotionally aroused an individual is by the visual stimuli, the more SCR is increased. SCR will be reported in microsiemens for each resting state period. Resting-state Electroencephalogram (EEG) will be recorded. EEG is measured in microvolts, refers to the spontaneous electrical activity in the brain during resting-state (i.e., no task).
Number of participants who had higher event-related potentials (ERPs) in response to CS+ categories relative to CS- categories, as assessed by electroencephalogram (EEG) during the image familiarization phase (viewing phase) | During the image familiarization/viewing phase (about 15 minutes total)
  On day 1 during the image familiarization phase (also called the viewing phase), participants will be presented with images on a computer screen from three different object categories, such as fruits, animals, and tools, and participants will be instructed to passively view the presented images.
  During the viewing phase, event-related potentials (ERPs) will be recorded to assess participants' response to each object category. Event-related potential (ERP), which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli.
Number of participants who had higher event-related potentials (ERPs) in response to CS+ categories relative to CS- categories, as assessed by electroencephalogram (EEG) during the fear conditioning phase | During the image familiarization/viewing phase (about 15 minutes total)
  On day 1, after the viewing phase, participants will then complete the fear conditioning phase. Participants will continue to be presented with images from the three categories. During the fear conditioning phase, ERPs will be recorded to assess participants' response to each object category.ERP), which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli.
Number of participants who had higher event-related potentials (ERPs) in response to CS+ categories relative to CS- categories, as assessed by electroencephalogram (EEG) during the avoidance learning phase | During the avoidance learning phase (about 18 minutes total)
  On day 1, after the fear avoidance phase, participants will complete the avoidance learning phase. In this phase, participants can or can not avoid a shock by pressing a button.
  During the avoidance learning phase, ERPs will be recorded to assess participants' response to each object category. Event-evoked potential (EEP), which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli.
Number of participants who had higher event-related potentials (ERPs) in response to CS+ categories relative to CS- categories, as assessed by electroencephalogram (EEG) during the memory recall phase | During the memory recall phase (about 18 minutes total)
  On day 2, participants will complete the memory recall phase. During this phase, participants will again be presented with images on a computer screen from three different object categories, such as fruits, animals, and tools. Participants will be informed that they have a choice to press or not to press a button during the CS presentation to avoid a possible shock.
  During the memory recall phase, ERPs will be recorded to assess participants' response to each object category. ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli.
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately Before the Viewing Phase on day 1
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately After the Viewing Phase (day 1 about 15 minutes after start of viewing phase)
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately Before the fear conditioning Phase (day 1 about 20 minutes after start of viewing phase)
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately After the fear conditioning Phase (day 1 about 38 minutes after start of viewing phase)
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately Before the avoidance learning phase (day 1 about 43 minutes after start of viewing phase)
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately after the avoidance learning phase (day 1 about 61 minutes after start of viewing phase)
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately Before the memory recall phase on day 2 (about 1 day after start of viewing phase
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Spontaneous electrical activity in the brain during the resting state as assessed by electroencephalogram (EEG) | Immediately after the memory recall phase (day 2 about 1 day 18 minutes after start of memory recall phase).
  ERP, which is assessed by electroencephalogram (EEG) and measured in microvolts, refers to the electrical activity in the brain that is elicited by a specific stimuli. EEG will be recorded during the resting states immediately before and after each experimental phase (the 4 experimental phases are the viewing phase on day 1, the fear condition phase on day 1, the avoidance learning phase on day 1, and the memory recall phase on day 2).
Number of times a participant pressed the button to avoid shock in response to an object category during the avoidance learning phase | During the avoidance learning phase (about 18 minutes total)
  On day 1, after the fear avoidance phase, participants will complete the avoidance learning phase. In this phase, participants can or can not avoid a shock by pressing a button.
  During the avoidance Learning Phase, the number of time a participant presses the button in response to each of the 3 object categories will be reported.
Number of times a participant pressed the button in response to an object category during the memory recall phase | During the memory recall phase (about 18 minutes total)
  On day 2, participants will complete the memory recall phase. During this phase, participants will again be presented with images on a computer screen from three different object categories, such as fruits, animals, and tools. Participants will be informed that they have a choice to press or not to press a button during the CS presentation to avoid a possible shock.
  During the memory recall phase, the number of time a participant presses the button in response to each of the 3 object categories will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milad, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No